CLINICAL TRIAL: NCT05371457
Title: The Influences of Subscapularis Lesion on Ultrasonography and Scapular Kinematics in Patients With Shoulder Impingement Syndrome
Brief Title: The Influences of Subscapularis Lesion on Ultrasonography and Kinematics in Patients With Shoulder Impingement
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202011045RIND
Record Dates: First submitted 2022-02-06; First posted 2022-05-12 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2021-12

CONDITIONS: Shoulder Impingement Syndrome
Keywords: shoulder impingement syndrome; subcoracoid impingement; coracohumeral ligament distance; subscapularis
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Subacromial and subcoracoid impingement have been categorized as external impingement, one type of shoulder impingement syndrome (SIS). Differentiation between subacromial impingement and subcoracoid impingement are important in determining the treatment target. The thickness of the coracohumeral ligament (CHL) may affect coracohumeral distance (CHD), which has been suggested as a possible factor in developing subcoracoid impingement with subscapularis (SSC) lesion. Evidence that indicates the existence of abnormal SSC, CHL thickness and CHD in people with SIS is limited. The purposes of the study were (1) to evaluate the correlations between CHL thickness and CHD by using ultrasonography in people with SIS with and without SSC lesion, (2) to examine the difference in SSC/CHL thickness and CHD between people with SIS with and without SSC lesion.

DETAILED DESCRIPTION:
Based on previous studies, a total sample size of 40 participants was calculated to provide 80% power with detection of a difference of more than 1.0 mm CHD between 2 groups. The inclusion criteria of the participants were age of 20-60 years old and positive unilateral shoulder results on at least 3 of 5 tests: 1) Neer's test, 2) Hawkins' test, 3) the Empty can test, 4) the pain or weakness with resisted ER test, and 5) tenderness in the tendon of the rotator cuff. Participants with a history of shoulder dislocation, fracture or surgery, history of direct contact injury to the neck or upper extremities within the past month, glenohumeral joint instability (positive apprehension test, sulcus sign), neurologic disorder (upper motor neuron diseases, cervical radiculopathy), passive ER Range of Motion (ROM) less than 30 degrees, or pain (visual analogue scale, VAS more than 5) during the experimental tasks were excluded. After the impingement tests were performed to ensure that the participants met our inclusion criteria, all participants were assessed with 3 special SSC tests, namely, the lift-off test, belly-press test (Napoleon sign) and bear-hug test, for group allocation. Patients with positive results on at least 2 of the 3 special tests were allocated to the SSC lesion (SSCL) group.

The characteristics of the participants were collected by one assessor, including age, gender, height, weight, dominant side, involved side, duration of symptom, pain (VAS), occupation ratio, the Flexilevel Scale of Shoulder Function (FLEX-SF) and internal rotator strength.

USG measurements We measured the following outcomes: (1) CHL thickness, (2) CHD and (3) AHD. Each outcome was measured in 3 trials and the mean of the 3 trials was used for data analyses. All of the measurements were measured with THI turned on except for that of CHD, due to the deeper anatomical structure.

For measurement of the CHL thickness, the position of the linear probe was on the lateral border of the coracoid process to obtain a longitudinal image of the CHL. Each participant was instructed to lie in supine position and relax while the examiner maintained the elbow of the participant at flexion of 90° and the shoulder under maximal ER without shoulder abduction or flexion (arm by side) (Figure 2). Maximal ER of the shoulder was achieved when the examiner could not further externally rotate the shoulder of the participant. The thickness of the CHL at a 2-mm distance from the coracoid process was measured.

CHD was measured with the probe positioned on the lateral border of the coracoid process to obtain images of the coracoid process and humeral head in 4 different shoulder rotation positions: (1) shoulder neutral rotation (CHD-NR), (2) external rotation (CHD-ER) and (3) shoulder internal rotation with maximal forward flexion and full adduction (CHD-IRFA, with the arm adducted across the chest reaching for the opposite shoulder) and (4) shoulder internal rotation (CHD-IR) (Figure 2). Participants were asked to sit with their arms by their sides and to perform the 4 different positions respectively. The measurements were repeated for 3 trials with repositioning of the arm to a neutral position for intervals of 10 seconds. The distance measured was that between the coracoid process and the lesser tuberosity of the humerus.

SSP tendon thickness was evaluated with the patient's palm placed over his/her iliac wing, or "back pocket", with the elbow flexed and directed medially. The transducer was placed over the anterior aspect of the shoulder, perpendicular to the supraspinatus tendon and just anterior of the anterior-lateral margin of the acromion. A transverse glide was then performed at the site to determine the exact position where the observer judged that the tendon thickness was at its maximum. The thickness of the SSP tendon was measured 2 cm away from the biceps long head tendon. For measuring SSC tendon thickness with a short axis of view, the probe was positioned horizontally on the bicipital grove. The participant's forearm was placed with the elbow flexed to 90° in slight internal rotation, with the palm facing upward and medially. Then the patient was asked to rotate the forearm externally, keeping the palm up and the elbow strictly close to the iliac crest.

Acrociohumeral distance (AHD) was measured under 0° and 60° of scapular plane shoulder elevation. The transducer was placed on the most anterior aspect of the acromion edge, with the long axis of the transducer placed in the plane of the scapula and parallel to the flat surface of the acromion. The participants sat in an upright position without back support and with their feet flat on the floor, holding their shoulders back and looking straight ahead, to achieve retracted shoulders and extension in the thoracic and cervical spine. AHD was measured at 0° and 60° of active shoulder elevation in the scapular plane. A 60° scapular elevation of AHD was then measured with a goniometer placed on the patient's arm to determine 60° of active shoulder elevation, with the thumb pointing up.

ELIGIBILITY:
Inclusion criteria:

1. Age from 20 to 60 years old
2. Unilateral shoulder symptoms

2. At least three positive of five tests, including Neer's test, Hawkin's test, Empty can test, tenderness in tendon of rotator cuff and resisted external test.

Exclusion criteria:

1. Shoulder dislocation
2. Fracture
3. Surgery
4. History of direct contact injury to the neck or upper extremities within the past month
5. Glenohumeral joint instability (positive apprehension test, sulcus sign)
6. Neurologic disorder (upper motor neuron diseases, cervical radiculopathy)
7. Passive ER ROM less than 30 degrees
8. Pain (visual analogue scale, VAS more than 5)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Forty subjects whose age from 20 to 60 years old were recruited from National Taiwan University Hospital and through general local internet media. The inclusion criteria of subjects will be at least three positive of five tests, including Neer's test, Hawkin's test, Empty can test, tenderness in tendon of rotator cuff and resisted external test. In addition, participants with a history of shoulder dislocation, fracture or surgery, history of direct contact injury to the neck or upper extremities within the past month, glenohumeral joint instability (positive apprehension test, sulcus sign), neurologic disorder (upper motor neuron diseases, cervical radiculopathy), passive ER ROM less than 30 degrees and pain (visual analogue scale, VAS less than 5) during the experimental tasks will be excluded.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Thickness of Coracohumeral Ligament (CHL) | Baseline
  The T3300 ultrasound system (BenQ, Taipei, Taiwan) is a portable ultrasonography machine to collect thickness of CHL as well as CHD. B-mode US depicts the CHL as a linear hyperechoic band surrounded by hyperechoic fat. Differentiation of the CHL from surrounding tissues can be achieved by tilting the probe to show anisotropy and by dynamic examination IR and ER. The CHL will be loosened (concave) in IR and tightened (straight) in ER. During the maximal ER, the thickness of the CHL at a 2-mm distance from the coracoid process will be measured.
Coracohumeral Distance (CHD) | Baseline
  CHD was measured with the probe positioned on the lateral border of the coracoid process to obtain images of the coracoid process and humeral head in 4 different shoulder rotation positions: (1) shoulder neutral rotation (CHD-NR), (2) external rotation (CHD-ER) and (3) shoulder internal rotation with maximal forward flexion and full adduction (CHD-IRFA, with the arm adducted across the chest reaching for the opposite shoulder) and (4) shoulder internal rotation (CHD-IR). Participants were asked to sit with their arms by their sides and to perform the 4 different positions respectively. The measurements were repeated for 3 trials with repositioning of the arm to a neutral position for intervals of 10 seconds. The distance measured was that between the coracoid process and the lesser tuberosity of the humerus. The distance will be measured in the shortest distance between the interval of coracoid process and the lesser tuberosity of the humerus.
Long Head of Biceps Tendon (LHBT) Stability | Baseline
  dynamic stability assessment and presence of "chondral print" will be measured for LHBT stability. The probe will be placed at the level of bicipital groove and slightly move upward for short axis image (dynamic stability and "chondral print") and orientated perpendicularly between the bicipital groove for long axis image ("chondral print"). The participant's forearm is placed with the supinated elbow flexed 90° and 10° of IR. Then, the LHBT transposition will be recorded while asking the participant to externally and internally rotation of GH joint for dynamic stability assessment. For "chondral print" evaluation, investigate the presence of irregularity of bicipital groove under short and long axis view.
Humerus elevation | Baseline
  The Polhemus 3Space FASTRAK system (Polhemus Inc., Colchester, VT, USA) is an electromagnetic motion analysis system with Motion Monitor software which is used to collect three-dimensional scapular kinematics. The sensors will be attached to bony landmarks (sternum, the scapular acromial process, and the distal humerus between the lateral and medial epicondyles). The recording will be started with the participants in a sitting position, and two hands at the sides. Then, the participants will be asked to perform 5 trials of full ROM scapular plane elevation, and simultaneously we measuring the kinematic data. The humerus elevation, scapular upward/downward rotation, anterior/posterior tipping and internal/external rotation, elevation/depression will be calculated by the software. The kinematic data will be recorded during 30°, 60°, 90° and 120° in raising and lowering phase of humeral elevation in the scapular plane.
Scapular upward/downward rotation | Baseline
  See outcome 4
Scapular anterior/posterior tipping | Baseline
  See outcome 4
Scapular internal/external rotation | Baseline
  See outcome 4
Scapular elevation/depression | Baseline
  See outcome 4
Scapular muscles activities | Baseline
  Electromyography surface silver chloride circular electrodes with an interelectrode distance of 20 mm, and a Grass AC/DC amplifier with a gain of 1,000, a common mode rejection ratio of 86 dB at 60 Hz, and a bandwidth (-3 dB) of 10 - 1,000 Hz were used. The sEMG data will be collected at 2,000 Hz/channel using a 16-bit analog to digital converter. Each electrode will be controlled with an impedance less than 10 k. The procedures of the recording of the sEMG activity are the same as the kinematic data. A RMS algorithm will be used to produces sEMG envelopes with a sampling rate of 50. Results will be normalized to the maximal activity during MVIC trials. Upper trapezius(UT), long head of biceps(LHB), lower trapezius(LT) and serratus anterior(SA) muscle activation in 0-30°, 30°-60°, 60°-90°, 90°-120° and >120° in raising and lowering phase will be recorded. The mean sEMG amplitude of each phase will be reported as a percentage of MVIC to assess the activity of each muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Jiu- Jenq Lin, PHD, Principal Investigator — School and Graduate Institute of Physical Therapy College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan